CLINICAL TRIAL: NCT04907955
Title: Visual Performance Following Implantation of 3 Presbyopia Correcting Intraocuar Lenses
Brief Title: Visual Performance Following Implantation of Presbyopia Correcting IOLs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dar Al Shifa Hospital (Other)
Responsible Party: Principal Investigator, magda torky, Principle investigator, Dar Al Shifa Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02282021065727
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Loss of Visual Contrast Sensitivity; Near Vision; Visual Impairment
MeSH Terms: conditions — Myopia; Vision Disorders | interventions — Phacoemulsification

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- panoptix PANFOCAL intraocular lens (Active Comparator): panoptix PANFOCAL intraocular lensis a single-piece aspheric non-apodized diffractive panfocal IOL that distributes light energy to three focal points in both small and large pupil conditions
  Interventions: Procedure: phacoemulsification with implantation of presbyopia correcting IOL
- Trifocal Diffractive the AT LISA intraocular lens (Active Comparator): Trifocal Diffractive the AT LISA is a preloaded single-piece aspheric diffractive trifocal IOL and made of hydrophilic acrylic with a hydrophobic surface with an ultraviolet absorber. This aspheric IOL is aberration -correcting in order to reduce and compensate for corneal spherical aberrations.
  Interventions: Procedure: phacoemulsification with implantation of presbyopia correcting IOL
- Symphony EDOF (extended depth of focus) intraocular lens (Active Comparator): SYMPHONY EDOF intraocular lens is a single-piece aspheric biconvex hydrophobic acrylic IOL with a 6.0 mm optic and an 13.0 mm overall diameter. This IOL consists of a wavefront-designed anterior aspheric surface (negative spherical aberration of -0.27 mm to counterbalance the net positive spherical aberration from cornea) and a posterior achromatic diffractive surface with echelette design.
  Interventions: Procedure: phacoemulsification with implantation of presbyopia correcting IOL

INTERVENTIONS:
Procedure: phacoemulsification with implantation of presbyopia correcting IOL — cataract extraction with phacoemulsification and insertion of presbyopia correcting IOL

SUMMARY:
The purpose of the current study was to compare the visual performance after bilateral implantation of the Panoptix IOL , or the AT LISA IOL or Tecnis Symfony IOL . The focus was on intermediate vision, defocus curves, and contrast sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* patients with normal ocular examination apart from cataract.

Exclusion Criteria:

* previous ocular surgery.
* ocular pathology or corneal abnormalities.
* an endothelial cell count below 2000 cells/mm2.
* corneal astigmatism greater than 1.0 diopter (D) measured with Scheimpflug tomography (Sirius, CSO, Italy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
visual acuity | 6 months postoperatively.
  The monocular uncorrected (UDVA) and corrected (CDVA) distance visual acuity (4 m), uncorrected intermediate visual acuity (UIVA) (60 cm and 80 cm), distance-corrected intermediate visual acuity (DCIVA), uncorrected near visual acuity (40 cm), and distance-corrected near visual acuity (DCNVA) were assessed. Standardized logarithm of the minimum angle of resolution (logMAR) charts were used for visual acuity measurement at 4 m, 80 cm, and 40 cm.

SECONDARY OUTCOMES:
defocus curve | 6 months postoperatively.
  The binocular defocus curve was done to evaluate the functional range of vision. The curve was obtained while the patient wearing his distance correction to provide the best distance visual acuity in both eyes. The test was performed under photopic conditions (85 candelas/m2) using ETDRS charts at a distance of 4m with the introduction of defocusing lenses from +1.00 D to -4.00 D in 0.50 D steps.
contract senstivity | 6 months postoperatively.
  The CSV-1000 system (Vector Vision Inc. Greenville, OH, USA) was used to measure contrast sensitivity under photopic and mesopic conditions without glare with spatial frequencies ranging between 3 and 18 cycles/degree.
photic phenomena | 6 months postoperatively.
  The presence of dysphotopsia including haloes, glare and starburst were assessed regarding their frequency, severity and the degree of bother.
spectacle independence | 6 months postoperatively.
  patients were given a questionnaire to assess their spectacle independence. The response for spectacle independence was yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Daralshifa hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No